CLINICAL TRIAL: NCT02444273
Title: The Feasibility of a Prehabilitation Program in the Liver Transplant Population at Barnes-Jewish Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201403118
Record Dates: First submitted 2015-04-07; First posted 2015-05-14 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: End Stage Liver Disease; Physical Activity
Keywords: liver diseases; liver transplantation; preoperative care; physical therapy
MeSH Terms: conditions — End Stage Liver Disease; Motor Activity; Liver Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Subjects will receive standard care both pre and post transplant.
- Exercise Group (Experimental): Subjects will receive a personalized home exercise program and regular phone calls from a therapist to monitor and promote activity.
  Interventions: Procedure: Exercise

INTERVENTIONS:
Procedure: Exercise — Subjects will be given and individualized exercise program.
  Arms: Exercise Group

SUMMARY:
The primary outcome of this study is to demonstrate the feasibility of a prehabilitation program at Barnes Jewish Hospital for liver transplant candidates. Those patients who consent to participate in the study and are placed on the transplant list will be randomized into either the control or intervention group. The intervention group receives a personalized home exercise program along with weekly phone calls to provide coaching, mentoring and motivation. Data collected at baseline, post-transplant and, post-transplant follow up will be compared among the two study groups. The secondary outcomes include: normative data of functional measures for patients with end stage liver disease and to determine the effect size for future research on prehabilitation in the patient population.

ELIGIBILITY:
Inclusion Criteria:

* Being evaluated for liver transplantation by Barnes Jewish Hospital medical team

Exclusion Criteria:

* Non-english speaking
* Medical contraindications to exercise as determined by the medical team

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of a prehabilitation program. | 2 Years
  Feasibility will be measured by participation and outcome assessment measures.

SECONDARY OUTCOMES:
Normative data on Timed Up and Go for patients with end stage liver disease. | Baseline
Normative data on 10 meter walk for patients with end stage liver disease. | Baseline
Normative data on Modified Dynamic Gait Index for patients with end stage liver disease. | Baseline
Normative data on Five Time Sit to Stand for patients with end stage liver disease. | Baseline
Normative data on 6 Minute Walk Test for patients with end stage liver disease. | Baseline

IPD SHARING:
Plan to Share IPD: Undecided